CLINICAL TRIAL: NCT00783003
Title: A Single Centre, Randomised, Placebo-controlled, Four-way Cross Over Study to Assess the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Inhaled Doses of GSK233705 and GW642444 as Monotherapies and in Combination in Healthy Japanese Subjects
Brief Title: A Study to Assess the Safety and Pharmacokinetics of Inhaled Doses of GSK233705 and GW642444 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 112146
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Tolerability; Muscarinic Receptor Antagonist, Anticholinergic; Safety; Anticholinergic; ß2 agonist; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Long acting muscarinic receptor antagonist (LAMA) (Experimental): Inhaled Long acting muscarinic receptor antagonist (LAMA which is in development as a treatment for Chronic Obstructive Pulmonary Disease.
  Interventions: Drug: GSK233705
- Long acting Beta 2 agonist (LABA) (Experimental): Inhaled Long Acting Beta 2 agonist (LABA) which is in development as a treatment for Chronic Obstructive Pulmonary Disease.
  Interventions: Drug: GW642444
- LAMA with LABA (Experimental): Inhaled Long Acting Muscarinic receptor Antagonist (LAMA) and a inhaled Long Acting Beta 2 Agonist (LABA), both in development for treatment of Chronic Obstructive Pulmonary Disease and taken in combination.
  Interventions: Drug: GSK233705 and GW642444
- Placebo (Placebo Comparator): Matching placebo, no intervention.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GSK233705 and GW642444 — Inhaled Long acting muscarinic receptor antagonist (LAMA) and a inhaled Long acting Beta 2 agonist (LABA) both in development as treatment for Chronic Obstructive Pulmonary Disease, taken in combination.
  Arms: LAMA with LABA
Drug: GW642444 — Inhaled Long acting Beta 2 agonist (LABA)
  Arms: Long acting Beta 2 agonist (LABA)
Drug: GSK233705 — Inhaled Long acting muscarinic receptor antagonist (LAMA which is in development as a treatment for Chronic Obstructive Pulmonary Disease.
  Arms: Long acting muscarinic receptor antagonist (LAMA)
Drug: Placebo — Matching placebo.
  Arms: Placebo

SUMMARY:
GW642444 and GSK233705 are in development for treatment of Chronic Obstructive Pulmonary Disease. Development of these two inhaled drugs as a combination therapy would have potential for improved patient benefit as they both work through different mechanisms and the combined bronchodilatory effect might be additive. This study will look at the this combination, for the first time, in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Japanese ethnic origin (defined as having been born in Japan with four ethnic Japanese grandparents and able to speak Japanese)
* Male or female between 18 and 65 years of age.
* Female subjects must be of non childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* Male subjects must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 90 days post-last dose.
* Body weight > 45 kg and body mass index within the range of 18-28 kg/m2 inclusive.
* Average QTc(B) < 450 msec taken from triplicate assessments at screening.
* No clinically active and relevant abnormality on 12-lead ECG at screening or 24h Holter ECG.
* Normal spirometry (FEV1 ≥ 80% of predicted, FEV1/FVC ≥ 70%).
* Non-smokers (never smoked or not smoking for >6 months with <10 pack years history (Pack years = (cigarettes per day smoked/20) x number of years smoked))
* A signed and dated written informed consent is obtained from the subject
* The subject is capable of giving informed consent, which includes compliance with the requirements and restrictions listed in the consent form
* Available to complete the study

Exclusion Criteria:

* Any clinically important abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG (12-lead). 24hr Holter monitoring outside normal limits.
* A history of breathing problems (i.e. history of asthmatic symptomatology, unless asthma in childhood that has now resolved and no longer requires maintenance therapy which should not be an exclusion).
* A mean QTc(B) value at screening >450msec, or an ECG that is not suitable for QT measurements (e.g. LBBB or poorly defined termination of the T wave).
* A history of elevated resting blood pressure or a mean blood pressure higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 40-90 bpm at screening.
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates and benzodiazepines. The detection of drugs with a legitimate medical use would not necessarily be an exclusion to study participation. The detection of alcohol would not be an exclusion at screening but would need to be negative pre-dose and during the study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody (if determined by the local SOP's).
* History of high alcohol consumption within 3months of the study defined as: an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males), or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females). One unit is equivalent to a half-pint (220mL) of beer or 1 (25ml) measure of spirits or 1 glass (125ml) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, (except for simple analgesics eg paracetamol), including vitamins, herbal and dietary supplements (including St John's Wort (Hypericum)) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels indicative of smoking or history of regular use of tobacco- or nicotine-containing products prior to screening.
* The subject is unable to use the novel dry powder inhaler correctly.
* The subject has a known allergy or hypersensitivity to ipratropium bromide, Tiotropium, atropine and any of its derivatives.
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug,
* The subject has a known allergy or hypersensitivity to milk protein or the excipients lactose monohydrate and MgSt.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-11-10 (Actual); Primary Completion 2009-02-06 (Actual); Study Completion 2009-02-06 (Actual)

PRIMARY OUTCOMES:
Heart rate | 24 hours
Systolic and diastolic blood pressure | 24 hours
12 lead ECG | 24 hours
Lung Function | 24 hours
Clinical laboratory safety tests | 24 hours
Adverse events | Duration of study

SECONDARY OUTCOMES:
Plasma concentrations of GSK233705 and derived pharmacokinetic parameters. | 24 hours
Plasma concentrations of GW642444 and derived pharmacokinetic parameters. | 24 hours
Weighted mean and minimum value potassium | 0 to 4 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Stepney Green, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 112146 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/112146?search=study&search_terms=112146#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112146 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register